CLINICAL TRIAL: NCT01707368
Title: Course of Psoriasis During Long Term Treatment With Calcipotriol Plus Betamethasone in Gel Formulation
Brief Title: Non-interventional Study of Long-term Treatment of Psoriasis With Calcipotriol Plus Betamethasone in Gel Formulation
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-Daivobet-longterm-NIS-2012
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-01

CONDITIONS: Psoriasis Vulgaris; Plaque Psoriasis
Keywords: Psoriasis; Psoriasis vulgaris; Plaque Psoriasis; Daivobet® Gel; Germany
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all eligible patients: Daivobet® Gel once daily on areas with plaque psoriasis, treatment duration up to 8 weeks for body skin areas except scalp (scalp up to 4 weeks), treatment may be repeated under medical surveillance.
  Interventions: Drug: Daivobet® Gel

INTERVENTIONS:
Drug: Daivobet® Gel — Once daily on areas with plaque psoriasis, treatment duration up to 8 weeks for body skin areas except scalp (scalp up to 4 weeks), treatment may be repeated under medical surveillance.

SUMMARY:
The purpose of this observational study is to document the course of disease and relapse management during treatment with Daivobet® Gel under consideration of patient's individual application habits under daily use conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with light to moderate psoriasis vulgaris of trunk and extremities and treatment with Daivobet® Gel was planned anyway.
* Minimum of 3 years diagnosed psoriasis vulgaris.

Exclusion Criteria:

* Previous therapy with Daivobet® Gel
* Systemic therapy of psoriasis vulgaris
* Contraindications of Daivobet® Gel in the German package insert
* people that are incapable to give free consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Psoriasis vulgaris visiting their attending dermatologist in the primary care clinic
Sampling Method: Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rosenberg, PD Dr. med., Principal Investigator — private practise, D- 49078 Osnabrück, Germany
Locations (1):
- PD Dr. med. Rosenbach, Osnabrück, Lower Saxony, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany between 8th September 2011 (retrospective data) and 15th May 2014. The planned observation period for each patient was about 12 months.
  The total planned sample size of this NIS was 1000 (analysable 750) patients.
Period: Overall Study
Arm/Group | All Eligible Patients
Started | 561
Completed | 393
Not Completed | 168

BASELINE CHARACTERISTICS:
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 561
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.05 (16.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283
  Male | 278
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 561
Affected body surface area (BSA) at admission [Count of Participants; unit: Participants]
  <2% | 45
  2-4% | 119
  4-6% | 138
  6-8% | 125
  8-10% | 83
  >10% | 51

OUTCOME MEASURES:

1. Primary Outcome: The Course of Disease and Relapse Management During Treatment With Daivobet® Gel Under Consideration of Patient's Individual Application Habits Under Daily Use Conditions.
Description: Number of exacerbations and relapses during one year observation time
Time Frame: 1 year
Population: Participants with at least one observation after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 529
Participants
  No relapse | 277
  1 relapse | 121
  2 relapses | 59
  3 relapses | 24
  More than 3 relapses | 48

2. Secondary Outcome: PGA (Physician's Global Assessment of Psoriasis Vulgaris Severity)
Description: 6--point verbal rating scale
Time Frame: Baseline
Population: Participants with at least one severity assessment after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 528
Participants
  Free of symptoms | 0
  Almost free of symptoms | 5
  Mild | 108
  Moderate | 350
  Severe | 60
  Very severe | 5

3. Secondary Outcome: PGA (Physician's Global Assessment of Psoriasis Vulgaris Severity)
Description: Assessment on 6-step scale from "no visible disease (O)" to "very severe disease (5)
Time Frame: 1 year
Population: Participants with at least one observation after baseline (last observation carried forward)
Measure: Count of Participants; unit: Participants
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 528
Participants
  Free of symptoms | 66
  Almost free of symptoms | 177
  Symptoms mild | 153
  Symptoms moderate | 115
  Symptoms severe | 16
  Symptoms very severe | 1

4. Secondary Outcome: Side Effects
Description: Number of participants with serious and non-serious adverse drug reactions.
Time Frame: 1 year
Population: All enrolled
Measure: Number; unit: Number of events recorded
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 561
Number of events recorded
  Serious with causal relation probable | 0
  Serious with causal relation possible | 0
  Serious, not related | 2
  Serious, causality not assessible | 1
  Non-serious, causal relation probable | 8
  Non-serious, causal relation possible | 5
  Non-serious, not related | 17
  Non-serious, causality not assessible | 29

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | All Eligible Patients
All-Cause Mortality (participants affected / at risk) | 2/561
Serious Adverse Events (participants affected / at risk) | 3/561
Other Adverse Events (participants affected / at risk) | 50/561
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Eligible Patients (N=561)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sudden death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Eligible Patients (N=561)
Drug ineffective (General disorders) | 42 (42)
Psoriasis (Skin and subcutaneous tissue disorders) | 5 (5)
Application site pustules (Infections and infestations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Sense of oppression (General disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Follikulitis (Infections and infestations) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Application site dryness (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Mean duration of observation per patients: Mean (SD): 40.47 (17.60) weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No